CLINICAL TRIAL: NCT00629941
Title: A Multi-Center, Open-Label Study Evaluating the Cytokine and Eyelid Margin Bacterial Load Levels of Subjects Diagnosed With Chronic Blepharitis Following Dosing With AzaSite® (Azithromycin Ophthalmic Solution) 1%
Brief Title: Safety and Efficacy Study of AzaSite® in Subjects With Blepharitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Inspire Pharmaceuticals, Inc., sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 041-104; P08652
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis | interventions — Azithromycin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AzaSite®

INTERVENTIONS:
Drug: AzaSite® — Ophthalmic solution; 1 drop in each eye BID for two days, then 1 drop in each eye QD for ~26 days

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of AzaSite® ophthalmic solution, 1% on signs & symptoms of blepharitis and tear cytokine and eyelid bacterial load levels

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe chronic blepharitis
* If female of childbearing potential, are non-pregnant and non-lactating

Exclusion Criteria:

* Had ocular surface surgery (LASIK, refractive, etc.) within the past year
* Unwilling to discontinue use of contact lenses during the study
* Have glaucoma
* Unable or unwilling to withhold the use of lid scrubs during the study
* Have a serious systemic disease or uncontrolled medical condition that in the judgment of the investigator could confound study assessments or limit compliance
* Currently using any preserved topical ocular medications (with the exception of unpreserved tear substitutes) at the time of entry into the study or during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change in clinical signs and symptoms associated with blepharitis | 8 weeks

SECONDARY OUTCOMES:
Standard ocular safety assessments | 4 weeks
Change in tear cytokine and eyelid bacterial load levels | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, MD, Study Director — Sponsor GmbH
Locations (2):
- United States (2):
  - Central Maine Eye Care, Lewiston, Maine
  - Ophthalmic Research Associates, Andover, Massachusetts